CLINICAL TRIAL: NCT06415019
Title: A Randomized, Controlled Study to Evaluate the Sensitizing Potential of BAY H006689, Naproxen 10% Topical Gel in Healthy Subjects Using a Repeat Insult Patch Test Design
Brief Title: A Study to Learn About Whether BAY H006689 Causes an Allergic Reaction When Applied as a Topical Gel in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 22640
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Pain; Healthy Volunteers
MeSH Terms: conditions — Pain | interventions — Naproxen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The treatments (IPs and control) will not be blinded to investigative personnel involved in the preparation/application and removal of treatments. However, the Investigator and trained evaluator involved in the evaluation of responses, will remain blinded during the course of the study until Database Lock and finalization of the Statistical Analysis Plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BAYHO06689 (Experimental): Topical application of BAYH006689 naproxen 10% topical gel on the intact skin
  Interventions: Drug: Naproxen (BAYH006689)
- Placebo (Placebo Comparator): Topical application of placebo gel which contains 0% of naproxen on the intact skin
  Interventions: Drug: Placebo Gel
- Negative control (Placebo Comparator): Topical application of the sterile 0.9% saline (negative control) on the intact skin
  Interventions: Drug: A solution of 0.9% Saline

INTERVENTIONS:
Drug: Naproxen (BAYH006689) — BAYH006689 gel will be dispensed directly on the patch
  Arms: BAYHO06689
Drug: Placebo Gel — Placebo gel will be dispensed directly on the patch
  Arms: Placebo
Drug: A solution of 0.9% Saline — 0.9% Saline will be dispensed directly on the patch.
  Arms: Negative control

SUMMARY:
Researchers are looking for a better way to treat muscle and joint pain. Researchers have seen that medicines which help reduce pain and inflammation could be safer when applied directly to the skin, called topical application, than when taken by mouth. However, recent studies have found that using these medicines on the skin can sometimes cause skin reactions such as redness, itching, or irritation in the area where the medicine is applied. However, reports of more serious side effects, affecting the entire body, from using these topical medicines are uncommon.

The study treatment BAYH006689 is under development to treat muscle and joint pain.

In this study, participants will be healthy and will not benefit from BAYH006689. However, the study will provide information on how to test BAYH006689 in future studies in people with muscle and joint pain.

The main purpose of this study is to check if BAYH006689 topical gel causes any skin reactions in healthy participants. The skin reactions will be assessed using a scale. This scale will provide scores for redness, swelling, and other signs of skin irritation.

In this study, researchers will randomly assign 3 sites, adjacent to each other, on the back of participants' bodies just below the shoulder blades.

The following gels will be applied 10 times at these sites as a patch three times a week for 21 days and once after 14-17 days:

* BAYH006689
* Placebo, which looks like the study drug but does not have any medicine in it.
* 0.9 % saline

Each participant will be in the study for around 6 to 8 weeks. During this time they will:

* receive assigned treatment gels at the identified skin sites
* have their skin reaction symptoms assessed

During the study, the doctors and their study team will:

* check the medical history of the participants
* check participants' health by performing urine tests
* ask the participants questions about how they are feeling and what adverse events they are having An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective of whether they think they are related or not to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Is 18 years of age or older
* Free of any systemic or dermatological disorder that may interfere with results or increase risk of adverse events (AEs)

Exclusion Criteria:

* Has a condition and/or is using medications that may interfere with the study results
* Pregnant or planning to get pregnant or breastfeeding
* Is currently participating in any clinical testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Skin sensitization potential | Up to 12 weeks
  Skin sensitization will be based on specific scoring criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22640